CLINICAL TRIAL: NCT01294228
Title: Rapid Evaluation of Acute Kidney Injury With NGAL in Acutely Ill Patients in the ICU
Acronym: REAL-ICU
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Sponsor
Other Study IDs: BSTE-0409
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center, prospective, observational study of patients that are admitted to the intensive care unit (ICU). This study does not include any treatment or intervention and it is considered Nonsignificant Risk.

DETAILED DESCRIPTION:
The study will be conducted in two phases. Phase One is specimen acquisition and subject diagnosis adjudication. Phase Two is biomarker testing.

Phase One

Approximately 850 adults admitted to general ICUs will be enrolled within 12 hours of receipt of ICU admission orders. Study specific whole blood and urine specimens will be collected.

There is an Adjudication Committee for this study. This committee is comprised of qualified, board-certified nephrologists.

Phase Two

During Phase Two, the plasma specimens will be divided amongst three clinical sites representative of the intended end users of this assay, and tested under a separate testing protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 21 years of age or older.
* Subjects must be admitted to an Intensive Care Unit (medical or surgical) and must be enrolled into this study within 12 hours of receipt of ICU admission orders.
* Subjects must be assessed as likely to be alive in the ICU for a minimum of 48 hours after enrollment.
* The following plasma/serum creatinine values must be available:
* Subjects that are admitted to the ICU following an elective surgery or procedure must have at least one pre-surgical/ pre-procedure creatinine value obtained in the 7 days prior to presentation to the ICU.
* Subjects that are admitted to the ICU for any reason other than following an elective surgery or procedure must have at least one creatinine value obtained greater than 7 days and up to 6 months prior to presentation to the ICU.

Exclusion Criteria

* Subjects either receiving or in imminent need of Renal Replacement Therapy.
* Subjects with evidence of chronic kidney disease stages 4 and 5 as evidenced by a pre-enrollment estimated GFR of less than 30 mL/min/1.73M2 (according to the 4-variable MDRD22).
* Subjects with any obstructive uropathy at the time of presentation to the ICU.
* Subjects with any known urothelial, urological or kidney malignancies.
* Subjects that have had any urologic procedure or surgery immediately prior to admission to the ICU.
* Subjects that have had any renal transplant or nephrectomy.
* Subjects that have had cardiovascular surgery involving cardiopulmonary bypass within the previous 7 days.
* Subjects that have participated in an interventional clinical study within the previous 30 days including studies with any investigational and non-investigational drugs.
* The inability to obtain written Informed Consent from the subject or an authorized representative.
* Subjects that have been previously enrolled in this study during a prior admission to the ICU.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All comers ordered to be admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Kellum, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (28):
- United States (25):
  - LA County / USC Medical Center, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - UC San Francisco General Hospital, San Francisco, California
  - St. Francis Sleep Allergy and Lungs, Clearwater, Florida
  - Queen's Medical Center, Honolulu, Hawaii
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - International Heart Institute of Montana, Missoula, Montana
  - Cooper University Hospital, Camden, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Mount Sinai Hospital, New York, New York
  - SUNY Stony Brook University Hospital, Stony Brook, New York
  - East Carolina University, Greenville, North Carolina
  - University Hospitals, Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Providence Regional Medical Center, Everett, Washington
  - Swedish Medical Center, Seattle, Washington
- Canada (3):
  - Vancouver Coastal Health, Vancouver, British Columbia
  - St. Boniface Hospital, Winnepeg, Manitoba
  - Capitol District Health Authority, Halifax, Nova Scotia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Clinical Study Population: All study participants underwent the same study procedures and their clinical data was analyzed as a homogenous population.
Period: Overall Study
Arm/Group | Clinical Study Population
Started | 1001
Completed | 1001
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants whom received an adjudicated diagnosis of either AKI or non-AKI.
Arm/Group | Clinical Study Population
Number analyzed (Participants) | 871
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (15.7)
Gender [Count of Participants; unit: Participants]
  Female | 375
  Male | 496
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62
  Not Hispanic or Latino | 809
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 16
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 187
  White | 625
  More than one race | 0
  Unknown or Not Reported | 12
Region of Enrollment [Number; unit: participants]
  Canada | 81
  United States | 790

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy of the Triage Neutraphil-Gelatinase Associated Lipocalin (NGAL) Test as an Aid in the Diagnosis of Acute Kidney Injury (AKI) in an All-comers ICU Setting.
Description: The efficacy of the Triage Neutraphil-Gelatinase Associated Lipocalin (NGAL) Test as an aid in the diagnosis of acute kidney injury (AKI) in an all-comers ICU setting. Final AKI diagnoses were established by an adjudication committee.
Time Frame: Prior to or within 72 hours.
Population: Study participants who had both an adjudicated AKI diagnosis and an evaluable T=0 (study enrollment) blood collection and associated test results.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Clinical Study Population
Number analyzed (Participants) | 782
Probability | 0.671 [0.609 to 0.733]

ADVERSE EVENTS:
Time Frame: 30 Days
Arm/Group | Clinical Study Population
Serious Adverse Events (participants affected / at risk) | 0/1001
Other Adverse Events (participants affected / at risk) | 0/1001

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days